CLINICAL TRIAL: NCT01451736
Title: Clinical and Cognitive Effects of Paliperidone Palmitate vs. Oral Risperidone in First-Episode Schizophrenia
Brief Title: Oral Risperidone Versus Injectable Paliperidone Palmitate for Treating First-Episode Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Keith Nuechterlein, Ph.D., Professor, Semel Institute for Neuroscience and Human Behavior, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P50 MH066286 Phase II; P50MH066286 (NIH); R092670SCH4005 (Other: Ortho-McNeil Janssen Scientific Affairs, LLC.); NCT01458379 (obsolete NCT alias)
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia (Recent-onset)
Keywords: First-episode Schizophrenia; Schizoaffective Disorder, Depressed Type (recent-onset); Schizophreniform Disorder; oral risperidone; long-acting injectable paliperidone palmitate; functional outcome
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Paliperidone Palmitate; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- paliperidone palmitate (Invega Sustenna) (Experimental): Participants will be provided paliperidone palmitate (Invega Sustenna), administered in injectible long-acting form, plus group skills training and case management
  Interventions: Drug: paliperidone palmitate
- oral risperidone (Active Comparator): Participants will be provided oral risperidone, plus group skills training and case management
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: paliperidone palmitate — long-acting injectable
  Other Names: Invega Sustenna
  Arms: paliperidone palmitate (Invega Sustenna)
Drug: risperidone — oral
  Other Names: Risperdal
  Arms: oral risperidone

SUMMARY:
This study will determine the efficacy of oral risperidone (Risperdal) versus long-acting injectable paliperidone palmitate (Invega Sustenna) in treating people with first-episode schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a severely disabling brain disorder. People with schizophrenia often experience hallucinations, delusions, thought disorders, and movement disorders. Proper treatment of first-episode schizophrenia may increase the chances of controlling disease progression on a long-term basis. People experiencing their first episode of schizophrenia are more responsive to treatment than those with chronic schizophrenia, but are also more susceptible to adverse treatment side effects. Atypical antipsychotic medications have been shown to produce fewer extrapyramidal side effects than older "typical" antipsychotics. Oral risperidone is an atypical antipsychotic medication that is very commonly used to control the symptoms of schizophrenia. Adherence to prescribed oral medication continues to be a major clinical issue. This study will determine the effectiveness of oral risperidone versus a long-acting injectible alternative, paliperidone palmitate, in treating people with first-episode schizophrenia. Impact on clinical symptoms and cognitive functioning will be examined.

Participants in this open label study will be randomly assigned to receive either orally administered risperidone or long-acting paliperidone palmitate administered via injection. Participants assigned to oral risperidone will receive medication in doses that are determined to be optimal by the study psychiatrist. Participants assigned to long-acting risperidone will receive an injection of paliperidone palmitate once every 4 weeks. Dosages will be adjusted as necessary to achieve the optimal dosage. Following 2 to 3 months to achieve outpatient oral risperidone dosage stabilization, the randomized medication conditions will begin and participants will be monitored for 1 year. Study visits will occur once weekly throughout the study. They will include psychiatrist monitoring of medication response and side effects; group therapy meetings focused on everyday living skills; family education about schizophrenia; and individual meetings with a case manager for counseling and evaluations of schizophrenia symptoms, work recovery, and social functioning.

ELIGIBILITY:
Inclusion Criteria:

1. A first episode of a psychotic illness is occurring or did occur within the last 2 years;
2. A diagnosis by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition(DSM-IV)of schizophrenia, schizoaffective disorder, depressed type, or schizophreniform disorder; and
3. Between 18 and 45 years of age.

Exclusion Criteria:

1. Neurological disorder (e.g., epilepsy) or significant head injury;
2. Significant alcohol or substance use disorder within the six months prior to the first episode and evidence that substance abuse triggered the psychotic episode or makes the schizophrenia diagnosis ambiguous;
3. Mental retardation, i.e. premorbid intelligence quotient (IQ) less than 70;
4. Insufficient acculturation and fluency in the English language to avoid invalidating research measures of thought, language, and speech disorder or of verbal abilities;
5. Residence likely to be outside of commuting distance of the University of California, Los Angeles (UCLA) Aftercare Research Program; or
6. Patient has shown an inadequate response to an adequate previous trial of oral or long-acting injectable risperidone, paliperidone, or paliperidone palmitate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2011-10; Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Exacerbation or relapse of psychotic symptoms | Evaluated for 12 months
  Exacerbation or relapse of psychotic symptoms, as measured by the Brief Psychiatric Rating Scale (BPRS)
Cognitive functioning based on Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery | Baseline to 12 months
  The Overall Composite Score from the MATRICS Consensus Cognitive Battery will be the primary cognitive outcome measure.
Role Functioning | Baseline to 12 months
  Role Functioning Scale (RFS; Goodman et al. 1993).

SECONDARY OUTCOMES:
Cognitive performance on test battery (MCCB) | Measured at baseline and 12 months
  The cognitive domain scores from the MATRICS Consensus Cognitive Battery (MCCB) will be used as secondary measures to identify the domains in which treatment effects occurred.
Insight (Awareness of Mental Disorder) | Measured at baseline and 12 months
  Awareness of illness, as assessed by the Scale to Assess Unawareness of Mental Disorder, Revised Version (SUMD-R)
Retention in treatment | Measured at 12 months
  Retention in treatment
Social functioning | Baseline to 12 months
  Social Functioning Scale (Goodman et al., 1993)
Emotional reactivity on psychophysiological measures | Measured at baseline and 12 months
  Emotional reactivity on psychophysiological measures

CONTACTS AND LOCATIONS:
Overall Officials: Keith H Nuechterlein, Ph.D., Principal Investigator — University of California, Los Angeles (UCLA) Semel Institute for Neuroscience and Human Behavior
Locations (1):
- UCLA Semel Institute for Neuroscience and Human Behavior, Los Angeles, California, United States